CLINICAL TRIAL: NCT05351736
Title: Impact of Structural and Myelin Abnormalities on Cognitive Impairments in Recent-onset Schizophrenia - Before and After Lurasidone Treatment (MARYLU)
Acronym: MARYLU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-003816-20
Record Dates: First submitted 2022-02-24; First posted 2022-04-28 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Recent-onset schizophrenia (Experimental): Patients diagnosed with schizophrenia with onset in the last 5 years that will be started on lurasidone or that have been on treatment with lurasidone for less than two weeks at the time of enrollment.
  Interventions: Drug: Lurasidone

INTERVENTIONS:
Drug: Lurasidone — Treatment with lurasidone

SUMMARY:
The present longitudinal study aims to investigate the impact of lurasidone treatment in recent-onset psychosis patients. The effects of lurasidone will be studied primarily in terms of structural and myelin modifications, in relation to clinical outcomes, before and after treatment and in healthy controls. Furthermore, neuropsychological tests will be used to evaluate changes in cognitive performance.

ELIGIBILITY:
Inclusion Criteria for the experimental arm:

* Patients diagnosed with schizophrenia with onset in the past 5 years, diagnosed through a structured clinical interview (SCID-5 CV)
* Aged between 18 and 35 years
* Patients requiring treatment with lurasidone (independently from the inclusion in the present study) or that are being treated with lurasidone for 2 weeks maximum.
* no other psychotropic treatment during the 2 weeks preceding the beginning of the study
* Acceptance of the informed consent form for the participation to the study
* For women in childbearing age, negative pregnancy test (urine or blood Beta HCG) performed before the start of the treatment and use of a highly efficient contraceptive method (such as progestin contraceptives, estrogen-progestin contraceptives, IUD, IUS, bilateral fallopian tube blockage, vasectomized partner, sexual abstinence) throughout the duration of the treatment.

Exclusion Criteria for the experimental arm:

* presence of other psychiatric and/or neurological diagnoses
* previous antipsychotic treatment, except for patients that have been treated with other antipsychotics for less than a month and that have not been treated in the two weeks preceding the beginning of the trial, who are considered eligible.
* contraindications to lurasidone treatment (as per summary of product characteristics)
* intellectual disability
* alcool or substance abuse in the previous 6 months
* presence of absolute or relative contraindications to MRI
* underage patients
* no negative pregnancy test or no use of a highly efficient contraceptive method
* pregnancy (if a patient becomes pregnant during the course of the study, the subject will be excluded from the study)

Inclusion criteria for healthy controls:

* Aged between 18 and 35 years
* Acceptance of the informed consent form for the participation to the study

Exclusion criteria for healthy controls:

* presence of psychiatric and/or neurological disorders
* family history of psychiatric disorders in 1st-degree relatives
* intellectual disability
* other medical conditions at the time of the study
* family history of hereditary neurological diseases
* alcool or substance abuse
* presence of absolute or relative contraindications to MRI
* underage patients
* no negative pregnancy test or no use of a highly efficient contraceptive method
* pregnancy (if a subject becomes pregnant during the course of the study, the subject will be excluded from the study)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2024-01-28 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
Changes in brain structural modifications in terms of grey matter volume measured using magnetic resonance imaging | Before and at three months of treatment
  Modifications of grey matter volume measuring using magnetic resonance imaging
Changes in brain structural modifications in terms of cortical superficial area measured using magnetic resonance imaging | Before and at three months of treatment
  Modifications of cortical superficial area measuring using magnetic resonance imaging
Changes in brain structural modifications in terms of cerebral cortex thickness measuring using magnetic resonance imaging | Before and at three months of treatment
  Modifications of cerebral cortex thickness measuring using magnetic resonance imaging
Changes in myelin integrity measured using magnetic resonance imaging | Before and at three months of treatment
  Modifications of myelinization status measured in terms of myelin water fraction using magnetic resonance imaging

SECONDARY OUTCOMES:
Evaluation of efficacy as assessed by Positive and Negative Syndrome Scale (PANSS) | once per month during three months of treatment
  Evaluation of changes in Positive and Negative Syndrome Scale with respect to the baseline. The PANSS is a 30-items scale assessing positive, negative, and general psychopathology associated with schizophrenia. Symptom severity for each item is rated in a 7-poing scale (1=absent; 7=extreme).
Evaluation of efficacy as assessed by Brief Psychiatric Rating Scale (BPRS) | once per month during three months of treatment
  Evaluation of changes in Brief Psychiatric Rating Scale (BPRS) with respect to the baseline. The BPRS is a scale assesses the level of 18 symptom constructs such as hostility, suspiciousness, hallucination, and grandiosity. Each symptom construct ranges from 1 (not present) to 7 (extremely severe).
Number of Adverse effects | three months of treatment
  Number of severe and non severe adverse effects
Changes in cognitive performance as assessed by Brief Assessment of Cognition in Schizophrenia (BAC-S) | once per month during three months of treatment
  Changes in Brief Assessment of Cognition in Schizophrenia (BAC-S) neuropsychological test scores with respect to the baseline. BAC-S is an assessment tool of cognitive function in patients with schizophrenia.
Structural differences in patients at baseline vs healthy controls measured using magnetic resonance imaging | baseline
  Grey matter volume differences in patients at baseline vs healthy controls
Myelinization differences in patients at baseline vs healthy controls measured using magnetic resonance imaging | baseline
  Differences in terms of myelin water fraction in patients at baseline vs healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Brambilla, Professor, Principal Investigator — S. C. Psichiatria - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico
Locations (1):
- S.C. Psichiatria - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy, Italy